CLINICAL TRIAL: NCT00213603
Title: Endoscopic Follow-up of Low Grade Precancerous Bronchial Lesions in High Risk Patients (SELEPREBB1)
Brief Title: Follow-up Modalities of Low Grade Precancerous Bronchial Lesions
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2001/032/HP; PHRC French ministry of Health
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Precancerous Conditions; Thoracic Neoplasms
Keywords: precancerous lesions; Lung cancer; Follow-up; Randomized study; Autofluorescence endoscopy; precancerous conditions
MeSH Terms: conditions — Precancerous Conditions; Thoracic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchial biopsies (fixed samples)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this multicentric French randomized trial is to determine the best auto fluorescence bronchial endoscopic follow-up strategy in high risk patients bearing low grade bronchial precancerous lesions. Subjects will be randomly assigned to one of the following arm :

(A) every 6 months clinical and chest Xrays follow-up without intermediate endoscopy, (B) every 6 months clinical and chest Xrays follow-up including repeated autofluorescence endoscopy and biopsies on a 6 months basis in case of low grade dysplasia or on a one year basis in patients without dysplasia.

After 36 months follow-up, each patient from the two groups will be subjected to a final autofluorescence endoscopy and biopsy and a Spiral Chest Xray.

The final analysis will compare between the two groups :

1. The probability of progression from an initially identified low grade lesion to a high grade lesion
2. The probability of respiratory epithelial tract progression assessed by the occurrence of a lung cancer or high grade lesion.
3. The characteristics of lung cancers detected in each arm
4. In both arm, the influence of risk factors and persistent exposure to tobacco on lesion evolutivity.

DETAILED DESCRIPTION:
The goal of this multicentric French randomized trial is to determine the best auto fluorescence bronchial endoscopic follow-up strategy in high risk patients bearing low grade bronchial precancerous lesions. This Trial compares two follow-up modalities : observation without endoscopy for a three year period (group A " light " follow-up), versus repeated autofluorescence endoscopies and biopsies every six months for three years (group B " intensive ").

Methods: 300 subjects at high risk for lung cancer will be included over a two year period and followed-up for three years. In each subject an auto-fluorescence endoscopy and a Chest CT scan will be performed before the enrollment into the trial. To be included the subject must present with an initial Chest CT scan not suspicious for lung cancer and bronchial biopsy showing a moderate dysplasia or a lower grade lesion.

Subjects will be randomly assigned to one of the following arm :

(A) every 6 months clinical and chest Xrays follow-up without intermediate endoscopy, (B) every 6 months clinical and chest Xrays follow-up including repeated autofluorescence endoscopy and biopsies on a 6 months basis in case of low grade dysplasia or on a one year basis in patients without dysplasia.

Stratifications factors for randomization are: Center, occupational exposure to respiratory carcinogens, presence of a bronchial low dysplastic lesion versus absence of dysplasia.

Bronchial biopsies samples will be centrally reviewed by a panel of Pathologists.

After 36 months follow-up, each patient from the two groups will be subjected to a final autofluorescence endoscopy and biopsy and a Spiral Chest Xray.

The final analysis will compare between the two groups :

1. The probability of progression from an initially identified low grade lesion to a high grade lesion
2. The probability of respiratory epithelial tract progression assessed by the occurrence of a lung cancer or high grade lesion.
3. The characteristics of lung cancers detected in each arm
4. In both arm, the influence of risk factors and persistent exposure to tobacco on lesion evolutivity.

First inclusion into the trial : July 2002, End of recruitment December 2005, End of follow- up : december 2008.

An ancillary study analysing the performances of fibered confocal fluorescence microscopy has been started in december 2005 after IRB/ethical comity approval. This ancillary study is only performed at the Rouen University Hospital Center.

ELIGIBILITY:
Inclusion Criteria:

* Patient with one or several of the following risk factor for lung cancer:

  * Tobacco consumption more than 30 pack years
  * Lung or ENT cancer history, cured
  * Occupational exposure to respiratory carcinogens
* Normal baseline CT scan
* Autofluorescence endoscopy showing moderate dysplasia or lower grade lesion
* Written informed consent

Exclusion Criteria:

* Treatment with Vit A derivative
* Contra indication for a fiberoptic bronchoscopy under local anesthesia.
* Known evolutive cancer
* Chest radiation therapy within 5 years before inclusion or chemotherapy within two years before inclusion.
* Impossibility for a 3 years follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects at high risks for developping a lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2002-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
occurence of high grade lesion or occurence of a cancer during endoscopic or clinical follow up | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Luc c Thiberville, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, Haute Normandie, France

REFERENCES:
- [Result] Thiberville L, Moreno-Swirc S, Vercauteren T, Peltier E, Cave C, Bourg Heckly G. In vivo imaging of the bronchial wall microstructure using fibered confocal fluorescence microscopy. Am J Respir Crit Care Med. 2007 Jan 1;175(1):22-31. doi: 10.1164/rccm.200605-684OC. Epub 2006 Oct 5. PMID 17023733
- [Derived] Guisier F, Deslee G, Birembaut P, Escarguel B, Chapel F, Bota S, Metayer J, Lachkar S, Capron F, Homasson JP, Taulelle M, Quintana M, Raspaud C, Messelet D, Benzaquen J, Hofman P, Baddredine J, Paris C, Cales V, Laurent P, Vignaud JM, Menard O, Copin MC, Ramon P, Bouchindhomme B, Tavernier JY, Quintin I, Quiot JJ, Galateau-Salle F, Zalcman G, Piton N, Thiberville L. Endoscopic follow-up of low-grade precancerous bronchial lesions in high-risk patients: long-term results of the SELEPREBB randomised multicentre trial. Eur Respir J. 2022 Sep 15;60(3):2101946. doi: 10.1183/13993003.01946-2021. Print 2022 Sep. PMID 35236723
- [Derived] Salaun M, Roussel F, Bourg-Heckly G, Vever-Bizet C, Dominique S, Genevois A, Jounieaux V, Zalcman G, Bergot E, Vergnon JM, Thiberville L. In vivo probe-based confocal laser endomicroscopy in amiodarone-related pneumonia. Eur Respir J. 2013 Dec;42(6):1646-58. doi: 10.1183/09031936.00191911. Epub 2012 Sep 27. PMID 23018901